CLINICAL TRIAL: NCT06664671
Title: The Effect of Thyme Oil on Asthma Control and Respiratory Parameters in Asthmatic Patients
Brief Title: The Effect of Thyme Oil in Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Associate Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024/126
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Asthma; Asthma Patients
Keywords: Asthma; thyme oil; Phytotherapy; Inspiration; Respiratory
MeSH Terms: conditions — Asthma; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Experimental
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): The product used, with NV-2016 code, contains Nature&Nurture thyme essential oil (10 µL) macra (Barcode No: 8697742121135, Registration No: 381751) and includes components such as 1,3 y-Terpinene, 2.7% p-Cymene, 5.6% linalool, 1.2% terpinen-4-ol, 1.2% borneol, 1.2% β-Bisabolene, 3.2% tymol, and 75.7% carvacrol. The thyme oil will be applied via an inhaler stick with patients instructed to inhale eight breaths, three times daily for four days.
  Interventions: Other: Experimental
- Placebo Group (Placebo Comparator): Patients will receive an empty inhaler stick with usage instructions, completing the same pre- and post-test procedures as the intervention group.
  Interventions: Other: Placebo
- Control (Other): Patients will complete pre- and post-test forms without any intervention.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Experimental — Patients will inhale thyme oil via inhaler sticks with instructions on proper usage, supervised by the researcher. Each patient will complete the Patient Introduction Form, Asthma Control Test, and pre-test sections of the Asthma Symptom and Respiratory Parameters Form. Measurements of FEV1 and FEV1/FVC will be recorded. On the fourth day of hospitalization, post-test data will be collected.
  Arms: Intervention Group
Other: Placebo — Patients will receive an empty inhaler stick with usage instructions, completing the same pre- and post-test procedures as the intervention group.
  Arms: Placebo Group
Other: Control (Standard treatment) — Patients will complete pre- and post-test forms without any intervention.
  Arms: Control

SUMMARY:
This study is a pre-test post-test randomized controlled trial aimed at examining the effects of thyme oil inhalation on asthma control and respiratory parameters in patients with asthma. It will be conducted with 150 patients (intervention group = 50, placebo group = 50, control group = 50) in the pulmonary ward of a Training and Research Hospital in eastern Turkey. Patients will use either thyme oil-infused or placebo inhaler sticks, inhaling for eight breaths, three times a day for four days. The placebo group will receive an empty inhaler stick, while no intervention will be applied to the control group. Data will be collected from November 2024 to February 2025. The effects of thyme oil will be measured using the Asthma Control Test, Asthma Symptom and Respiratory Parameters Form, FEV1 (Forced Expiratory Volume in 1 second), and FEV1/FVC (Forced Expiratory Volume in 1 second to Forced Vital Capacity ratio) (Modified Tiffeneau-Pinelli index) values.

Hypothesis: It is hypothesized that thyme oil inhalation will significantly improve respiratory function parameters and asthma control levels in patients with asthma.

DETAILED DESCRIPTION:
Aim of the Study This study aims to determine the effects of thyme oil on asthma control and respiratory parameters in patients with asthma.

Type of Study This study is a pre-test post-test randomized controlled experimental design.

Population The population comprises inpatients (N = 210) in the pulmonary ward of a Training and Research Hospital located in eastern Turkey. Based on a 95% confidence interval, 5% margin of error, and 95% power analysis, a minimum of 137 patients is required. To minimize attrition, the study aims to include 150 patients (intervention group = 50, placebo group = 50, control group = 50). Data will be collected between November 2024 and February 2025.

Intervention In this study, thyme oil aromatherapy will be applied via inhalation. The product used, with NV-2016 code, contains Nature&Nurture thyme essential oil (10 µL) macra (Barcode No: 8697742121135, Registration No: 381751) and includes components such as 1,3 y-Terpinene, 2.7% p-Cymene, 5.6% linalool, 1.2% terpinen-4-ol, 1.2% borneol, 1.2% β-Bisabolene, 3.2% tymol, and 75.7% carvacrol. The thyme oil will be applied via an inhaler stick with patients instructed to inhale eight breaths, three times daily for four days.

Data Collection Tools Data will be collected using the "Patient Introduction Form," "Asthma Control Test," and "Asthma Symptom and Respiratory Parameters Form."

* Patient Introduction Form: Created by researchers, this form includes 12 questions regarding age, weight, height, gender, marital status, education, employment, income, occupation, family asthma history, smoking, chronic illness, and asthma diagnosis duration.
* Asthma Control Test (ACT): Developed by Nathan et al and validated by Schatz et al, the ACT is suitable for assessing asthma in patients aged 12 years and older. The test includes five questions scored on a five-point Likert scale, assessing daytime and nighttime symptoms, rescue medication usage, and impact on daily activities over the past four weeks. Scores range from 5 to 25, with higher scores indicating better asthma control. ACT reliability in Turkish (Cronbach's alpha = 0.84) was established by Uysal et al.
* Asthma Symptom and Respiratory Parameters Form: This form was designed by researchers to assess symptoms (e.g., dyspnea, cough, chest wheezing) and includes FEV1 and FEV1/FVC respiratory parameters.

Data Collection Procedure Data collection will occur in a Teaching and Research Hospital's pulmonary ward from November 2024 to February 2025. Patients will be randomized into intervention, placebo, or control groups.

* Intervention Group: Patients will inhale thyme oil via inhaler sticks with instructions on proper usage, supervised by the researcher. Each patient will complete the Patient Introduction Form, Asthma Control Test, and pre-test sections of the Asthma Symptom and Respiratory Parameters Form. Measurements of FEV1 and FEV1/FVC will be recorded. On the fourth day of hospitalization, post-test data will be collected.
* Placebo Group: Patients will receive an empty inhaler stick with usage instructions, completing the same pre- and post-test procedures as the intervention group.
* Control Group: Patients will complete pre- and post-test forms without any intervention.

Data Analysis Data analysis will be conducted using SPSS. Shapiro-Wilk Test will assess normality. Significance is set at p < 0.05. If variables are normally distributed (p > 0.05), parametric tests will be applied. Chi-square analysis will be used for categorical data. Paired t-tests will assess within-group differences, while repeated-measures ANOVA will test differences across groups, with variance homogeneity and multivariate normality checks.

Ethics Ethical approval for the study was obtained from the Inonu University Clinical Research Ethics Committee, and institutional permission was granted by Batman Training and Research Hospital. The protocol follows the Helsinki Declaration, and all participants will be informed about data confidentiality, their right to withdraw, and that no charges or costs will be incurred.

Research Hypotheses

The following hypotheses will be tested regarding the effects of thyme oil:

* H1: Thyme oil is effective in alleviating or reducing the severity of asthma symptoms in patients with asthma.
* H2: Thyme oil improves respiratory parameters in patients with asthma.
* H3: Thyme oil enhances asthma control in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* - Patients admitted to the pulmonology ward with a diagnosis of asthma and expected to stay for at least 4 days,
* Patients admitted on their first day in the pulmonology ward,
* Age 18 or older,
* Alert and conscious,
* Open to communication and cooperation,
* Willing to participate in the study.

Exclusion Criteria:

* - Patients under 18 years of age,
* Patients with pregnancy,
* Patients with dementia and/or other organic mental disorders,
* Patients with any psychiatric diagnosis, and
* Patients who do not wish to participate in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Asthma symptoms | From enrollment to the end of treatment at 4 days
  Thyme oil effectively alleviates or reduces the severity of asthma symptoms in patients with asthma. Its influence on asthma symptoms is assessed through indicators such as shortness of breath, cough, nocturnal wheezing, chest wheezing, and secretions. The presence of these symptoms and their severity levels are determined using a 10 cm horizontal line scale, with one end labeled "None" and the other end labeled "Severe." This scale serves as a measurement criterion for the outcomes obtained from the study.
Respiratory parameters | From enrollment to the end of treatment at 4 days
  Thyme oil improves respiratory parameters in patients with asthma. Its influence on respiratory parameters is assessed using indicators such as FEV1/FVC and FEV1. These respiratory parameters are recorded in the asthma symptom form.
Asthma control | From enrollment to the end of treatment at 4 days
  Thyme oil enhances asthma control in patients with asthma, as measured by symptoms such as wheezing, coughing, shortness of breath, chest tightness or pain, frequency of nebulizer medication use, and interference with work. The maximum score for this assessment is 25, while the minimum is 5. The Asthma Control Test (ACT) scoring is categorized as follows: a score of 25 indicates "complete control," scores between 20-24 indicate "good control," and scores below 19 are classified as "uncontrolled." A higher score reflects better asthma control, whereas scores of 19 or below indicate that the condition is not well-managed, necessitating adjustments in treatment to achieve better control.
Respiratory parameters | From enrollment to the end of treatment at 4 days
  Thyme oil improves respiratory parameters in patients with asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- A patient in eastern Turkey, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the data of the research will be shared in international journals using English language.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Alavinezhad A, Hedayati M, Boskabady MH. The effect of Zataria multiflora and carvacrol on wheezing, FEV1 and plasma levels of nitrite in asthmatic patients. Avicenna J Phytomed. 2017 Nov-Dec;7(6):531-541. PMID 29299436
- [Background] Uysal MA, Mungan D, Yorgancioglu A, Yildiz F, Akgun M, Gemicioglu B, Turktas H; Turkish Asthma Control Test (TACT) Study Group. The validation of the Turkish version of Asthma Control Test. Qual Life Res. 2013 Sep;22(7):1773-9. doi: 10.1007/s11136-012-0309-1. Epub 2012 Nov 10. PMID 23143589
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908